CLINICAL TRIAL: NCT02115178
Title: Haemodynamic Effects During Anorectal Surgery in Spinal Anaesthesia With Low Dose Hyperbaric Bupivacaine : a Comparison of the Jack -Knife and Lithotomy Position
Brief Title: Haemodynamic Effects During Anorectal Surgery: a Comparison of the Jack -Knife and Lithotomy Position
Status: Completed | Type: Observational
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Jurgita Borodiciene, Ph Student, Lithuanian University of Health Sciences
Other Study IDs: LT22552; JUR2009 (Registry Identifier: JUR2009)
Record Dates: First submitted 2014-04-09; First posted 2014-04-15 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Anorectal Surgery Haemodynamic Changes
Keywords: Hemodynamic changes; Spinal anesthesia; Patient position; Impedance cardiography
MeSH Terms: interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lithotomy or Prone position
  Interventions: Other: Lithotomy or Prone position

INTERVENTIONS:
Other: Lithotomy or Prone position — The surgery, haemodynamic measurements will be performed in Lithotomy or Prone position

SUMMARY:
Background and Goal of Study: Minimal dose of spinal hyperbaric bupivacaine is commonly performed for adult anorectal surgery. This kind of anaesthesia can cause sinus bradycardia and hypotension wich reason is body position, autonomic nervus system reaction, reflex reaction even with low levels of sensory block. However, neither the publication of minimal doses of spinal hyperbaric bupivacaine effects of haemodynamic modifications nor their accuracy was widely discussed. The aim of the study is to make a comparison of the haemodynamic modifications due to minimal dose of spinal hyperbaric bupivacaine for adult anorectal surgery in lithotomy or jack knife position of steering impedance device.

Materials and Methods: Patients will be included which are over then 18 years old, who underwent anorectal surgery of the benign pathology, requiring spinal anaesthesia, were admitted in this clinical randomized study, hospitalized in Hospital of Lithuanian University of Health Sciences Kaunas Clinics and agree to participate to this study (written settlement). All patients were implicitly divided in to 4 groups by the position will be operating (lithotomy or jack knife position and by American Society of Anaesthesiologists (ASA) clas I-II and III-IV). Technique of anaesthesia were strictly standardized by protocol. All patients were premedicated with oral diazepam 5mg and diclofenac 100mg 60min before operation. After arrival in the operating theater peripheral vein 18 or 20G catheter was inserted, infusion therapy were started with crystalloid 5-7ml/kg/hour. Standard monitoring was used, including noninvasive arterial blood pressure (BP), electrocardiography (ECG), heart rate, peripheral oxygenation. Circulatory changes were recorded impedance device. 2 single-neck sensors connected vertically on both sides of the neck just below the ears lobe. Another pair of sensors attached on both sides of the chest processus xiphoid axillary line level. Thorax allows a variable electrical current, it travels through the lowest resistance (blood-filled aorta) and resistance is measured. For each heart contraction during changes in blood volume and velocity. Accordingly, replacing the resistors obtained by impedance settings.

Haemodynamic variables were recorded in patients in the use of impedance cardiograph:

1. arrives in the operating room;
2. seating on the operating table;
3. following the puncture;
4. 10 min after spinal puncture;
5. was laid in lithotomy or jack knife position;
6. in the beginning and the end of the operation;
7. patient was placed in the bed.

Each measurement was monitoring and recorded the following data( ar findings):

* Cardiac output (CO);
* Systemic vascular resistance (SVR);
* Systolic index (SI)
* Cardiac index (CI);
* Acceleration index (ACI);
* Heart rate (HR);
* Non-invasive systolic (SAP), diastolic (DAP) and mean (MAP) blood pressure;
* Peripheral oxygenation (SpO2); Patients were placed in the sitting position on the slab (operating table) back to the doctor. Dural puncture was made at L3-L4 or L4-L5 with 27G Tamanho spinal needle ( BBraun, Germany) by medial punction in aseptic condition, before the punction was injected lidocaine 1% subcutaneous. 0.5% 4mg of heavy bupivacaine and 0.01% 10µg fentanyl were injected over 2 minutes after free flow of cerebrospinal fluid was obtained. After sitting for 10 minutes ( sensory block was checked by the dermatomes with the methods of cold sensitivity) patients were asked to lie in the position wich operation will be done (lithotomy or jack knife position).

After 20 min. surgery was started. When anaesthesia was imperfect, 25-100µg of fentanyl was given IV. General anaesthesia will be give in case of failure . These cases will be value like a failure, patients will be exclude from the study.

Clinically significant hypotension will be define as a mean arterial blood pressure and heart rate decrease of 20% below baseline values. Systolic arterial blood pressure will reduce to 90mmHG limit, intravenous ephedrine 5-10 mg will be injected. If heart rate will reduce to 45 bpm, bradycardia will be treated with atropine 0,5 mg IV.

ELIGIBILITY:
Inclusion Criteria:

Adult patient ASA (American Society of Anaesthesiologists) I-IV Surgery in prone position or in lithotomy position Anorectal surgery

Exclusion Criteria:

* inability to give consent to inclusion in trial
* age less than 18 years
* the regional anaesthesia is contraindicated
* the overweight more then 30%
* taking psychotropic and painkillers to treat chronic diseases
* the movement of the patients body, including the shivering
* the patients height is the <120 or> 230 cm
* the patients body weight is <30 or> 155 kg.
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to department of surgery for minor anorectal surgery.
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2011-08; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Hemodynamic changes | During anaesthesia and surgery
  Hemodynamics measurements using non-invasive impedance cardiography device (BP, HR, SpO2, Cardiac Index, cardiac output, stroke volume, systemic vascular resistance)

CONTACTS AND LOCATIONS:
Overall Officials: Jurate Gudaityte, Assoc. Prof., Study Chair — Department of Anaesthesiology,Lithuanian University of Health Sciences
Locations (1):
- Department of Anesthesiology, Lithuanian University of Health Sciences, Kaunas, Lithuania

REFERENCES:
- [Derived] Borodiciene J, Gudaityte J, Macas A. Lithotomy versus jack-knife position on haemodynamic parameters assessed by impedance cardiography during anorectal surgery under low dose spinal anaesthesia: a randomized controlled trial. BMC Anesthesiol. 2015 May 6;15:74. doi: 10.1186/s12871-015-0055-3. PMID 25943374